CLINICAL TRIAL: NCT01374308
Title: Phase IIII Study of a Therapeutic Vaccine Candidate Containing Hepatitis B Virus (HBV) Core Antigen (HBcAg) and HBV Surface Antigen (HBsAg) for Treatment of Patients With Chronic HBV Infection
Brief Title: NASVAC Phase-III Trial in Chronic Hepatitis B (CHB) Patients
Acronym: NASVAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinical Research Organization, Dhaka, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NASVAC01
Record Dates: First submitted 2011-06-12; First posted 2011-06-15 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Hepatitis B
Keywords: NASVAC; Pegylated Interferon-2b; CHB
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NASVAC (Experimental): NASVAC will be administered every 2 weekly intra-nasally at a dose of 100 micro grams for 5 times followed by every 2 weekly administration of 100 micro grams intra-nasally plus 100 micro grams subcutaneously.
  Interventions: Biological: NASVAC
- Pegylated interferon alpha 2b (Active Comparator): Injection Pegylated interferon alpha 2b will be administered once weekly subcutaneously at a dose of 180 micro grams for 48 weeks
  Interventions: Drug: Pegylated interferon alpha 2b

INTERVENTIONS:
Biological: NASVAC — NASVAC will be administered every 2 weekly intra-nasally at a dose of 100 micro grams for 5 times followed by every 2 weekly administration of 100 micro grams intra-nasally plus 100 micro grams subcutaneously.
  Arms: NASVAC
Drug: Pegylated interferon alpha 2b — Injection Pegylated interferon alpha 2b will be administered once weekly subcutaneously at a dose of 180 micro grams for 48 weeks
  Other Names: Pegasys; Pegintron; Pegin; Optipeg; Peghebron
  Arms: Pegylated interferon alpha 2b

SUMMARY:
The general objective of the present clinical trial is to compare the therapeutic efficacy of a combination therapeutic vaccine containing hepatitis B surface antigen (HBsAg) and hepatitis B core antigen (HBcAg) [later called NASVAC] with a commonly used antiviral drug, pegylated interferon in patients with chronic hepatitis B (CHB).

DETAILED DESCRIPTION:
To collect and assess data on the therapeutic potential of the NASVAC in CHB patients regarding:

Reduction of the serum HBV DNA levels. Reduction in the levels of alanine aminotransferase (ALT) Clearance of hepatitis B e antigen (HBeAg) Negativation or lowering of HBsAg Anti-HBsAg/anti-HBeAg seroconversion

An additional objective of this study is to reconfirm the safety of NASVAC in CHB patients that has previously been shown by us in Phase I-II clinical trial in CHB patients.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg+ serology for more than 6 months before the beginning of the treatment.

In the last six months, according to HBeAg serostatus, for:

* HBeAg (-) patients, with a) baseline HBV DNA ≥ 103 and b) raised serum ALT (x >1 ULN) or significant hepatic necroinflammation and/or fibrosis (HAI-NI>4 and/or HAI-F >2) or liver stiffness >7.2 KPa.
* HBeAg (+) patients, with a) baseline HBV DNA ≥ 104 and b) and raised serum ALT (x >1.5 ULN) or significant hepatic necroinflammation and or fibrosis (HAI-NI>4 and/or HAI-F >2) or liver stiffness >7.2 KPa.
* Patients of both sex from 18 to 60 years-old
* No specific hepatitis B treatment at least for 6 months previous to the inclusion
* Voluntary signed informed consent to participate in the trial

Exclusion Criteria:

* Condition of HBV asymptomatic carrier or cirrhosis or patients with primary hepatocellular carcinoma
* Positive serological markers for hepatitis C
* Positive serological markers for HIV
* Previous specific anti-hepatitis B treatment in the last 6 months.
* Critically ill patient history of heart or renal failure, hypertension, hyperthyroidism, epilepsy, immunodeficiency diseases, malignancies or any non-controlled systemic disease.
* Pregnancy or nursing women. Women in fertile age without any contraceptive methods.
* Known severe allergic conditions (degree III or IV asthma, urticaria, dermatitis, bronchitis, etc. or hypersensitivity to any of the ingredients present in the preparation).
* Severe psychiatric dysfunction or another limitation that prevents the patient's consent.
* History of Autoimmune diseases (such as SLE, rheumatoid arthritis, multiple sclerosis, non controlled diabetes mellitus type 1)
* History of other hepatic diseases of different etiology (such as alcoholism, autoimmune hepatitis, drug induced hepatitis, Wilson's diseases, hemochromatosis)
* History of immune suppressive disorder or administration of immune suppressive-immune modulator drugs (including steroids) during or in the 6 months previous to the study.
* Very high transaminase levels at the beginning of treatment (ALT over 500 U/L) suggesting a not stable disease with risk for patient's health or acute flares over 15 times the upper limit of normality.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of study participants with virological and or biochemical response as a measure of efficacy | At week 96

CONTACTS AND LOCATIONS:
Overall Officials: Mamun A Mahtab, MSc MD FACG, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Farabi General Hospital, Dhaka, Bangladesh

REFERENCES:
- [Derived] Al Mahtab M, Akbar SMF, Aguilar JC, Guillen G, Penton E, Tuero A, Yoshida O, Hiasa Y, Onji M. Treatment of chronic hepatitis B naive patients with a therapeutic vaccine containing HBs and HBc antigens (a randomized, open and treatment controlled phase III clinical trial). PLoS One. 2018 Aug 22;13(8):e0201236. doi: 10.1371/journal.pone.0201236. eCollection 2018. PMID 30133478